CLINICAL TRIAL: NCT07159828
Title: A Phase 1 Open-label Study to Assess AXN-2510 Monotherapy in Adult Patients With Advanced Solid Tumors
Brief Title: A Study to Assess AXN-2510 Treatment in Adult Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Axion Bio, Inc (Industry)
Collaborators: Instil Bio (Industry)
Responsible Party: Sponsor
Organization: Instil Bio (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXN2510X2101
Record Dates: First submitted 2025-08-22; First posted 2025-09-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult
Keywords: PD-L1; VEGF; Immuno-Oncology; Solid Tumor; AXN-2510; IMM2510

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AXN-2510 (Experimental): AXN-2510 given as intravenous (IV) infusion every 3 weeks, for a maximum of 24 months of treatment or until discontinuation criteria is met. Two increasing dose levels will be tested.
  Interventions: Biological: AXN-2510

INTERVENTIONS:
Biological: AXN-2510 — AXN-2510 is an antibody with PD-L1 blocking and VEGF inhibition activity in one drug. This is called a bispecific antibody, because it has 2 activities. This immuno-oncology treatment is in development for the treatment of solid tumors. AXN-2510 is differentiated from other PD-L1 and VEGF bispecific antibodies by its ability to inhibit multiple VEGF molecules and also increased antibody-dependent cellular cytotoxicity (ADCC) that can directly kill PD-L1-positive tumor cells.

SUMMARY:
The goal of this clinical trial is to learn more about the side effects and best dose of AXN-2510 in adults with advanced solid tumors. The main questions it aims to answer are:

* What are the side effects of AXN-2510?
* Which is the best tolerated dose of AXN-2510?
* How long does AXN-2510 stay in your body?

Participants will receive AXN-2510 every 3 weeks. Participants will visit the clinic for checkups and tests several days during the first and third doses, and once every 3 weeks for other doses.

DETAILED DESCRIPTION:
This is a phase 1 study where all adult participants will receive AXN-2510. There will be 2 increasing doses of AXN-2510 given to participants, the dose given depends on when a participant enters the study. Next will be enrollment of 20 participants at the different doses to obtain more information about side effects, tolerability, and if the drug is helping.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of an advanced or metastatic solid tumor that is relapsed or refractory following previous therapy, and for which there is no available standard therapy.
* Availability of PD-L1 Tumor Proportion Score (TPS) or Combined Positive Score (CPS); OR willingness to submit tumor tissue, if available, for central testing.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Age ≥ 18 years at the time of signing the informed consent.
* Adequate hepatic function.
* Adequate renal function.
* Adequate bone marrow function.
* Adequate blood clotting function

Exclusion Criteria:

* Active, untreated brain metastases or leptomeningeal disease requiring immediate local therapy, with some exceptions.
* Concurrent malignancy that is progressing or requires active treatment, with some exceptions.
* Received prior treatment within 5 half-lives or 4 weeks prior to starting AXN-2510, whichever is shorter (6 weeks for nitrosourea or mitomycin-C). Patients with prostate or breast cancer may continue concurrent hormone therapy.
* Current use of immune-suppressive medication at the time of study enrollment, with some exceptions.
* Uncontrolled hypertension defined as blood pressure of ≥ 160 mmHg systolic and/or ≥ 95 mmHg diastolic.
* Gross hemoptysis within 2 months of enrollment (defined as coughing up ≥ 0.5 teaspoons of fresh blood or small blood clots).
* Concurrent use of therapeutic anticoagulation or anti-platelet agents.
* History of perforation and/or fistula of the gastrointestinal tract, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), acute gastrointestinal bleeding within 6 months before enrollment, or extensive bowel resection within 6 months prior to enrollment.
* History of stroke, transient ischemic attack, or clinically significant thromboembolic event within 6 months prior to enrollment.
* Tumors with radiographic evidence of blood vessel invasion, central necrosis or intratumor cavitation, encasement of organs (e.g. heart, trachea, esophagus, central bronchi) or major blood vessels (e.g. central pulmonary artery, central pulmonary veins, aorta, brachiocephalic artery, common carotid artery, subclavian artery, superior vena cava).
* Impaired cardiac function or significant diseases.
* History of pulmonary fibrosis or interstitial pneumonia, pneumoconiosis, chemical pneumonia, interstitial lung disease requiring steroids, or other diseases causing severe impairment of lung function.
* Unresolved toxicity higher than Grade 1 CTCAE v5 (or most current version) attributed to any prior therapy or procedure at Screening, with exceptions for alopecia or Grade 2 neuropathy.
* Any prior Grade 4 immune-mediated adverse event (imAE) or Grade 3 imAE requiring steroid treatment while receiving immunotherapy that has been documented within the 12 months prior to the enrollment period.
* Known human immunodeficiency virus (HIV) or acquired immune deficiency syndromes. Note: well-controlled HIV will be allowed.
* Positive hepatitis B surface antigen and/or hepatitis B core antibody (participants with negative polymerase chain reaction assay are permitted with appropriate antiviral therapy). If a hepatitis test was conducted and had a negative result within 30 days of enrollment, an additional test is not required at screening.
* Active hepatitis C infection with positive viral loads. Participants who have been treated for hepatitis C infection can be included if they have documented sustained virologic response of ≥ 12 weeks. If a hepatitis test was conducted and had a negative result within 30 days of enrollment, an additional test is not required at screening.
* Known history of any grade hypersensitivity reactions (despite appropriate premedication) to any known components of AXN-2510 or required premedication.
* Women who are pregnant or lactating.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that in the opinion of the investigator, might confound the results of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | The first cycle of treatment (Cycle 1, Days 1-21)
  A DLT is defined as a toxicity occurring during the DLT observation period
Incidence of adverse events (AEs) and serious adverse events (SAEs) | From the informed consent until Day 30 post-last dose.
  AEs are defined and graded according to the NCI CTCAE version 5.0

SECONDARY OUTCOMES:
Identify if AXN-2510 is helping patients. | Measured every 6 weeks for 48 weeks and every 12 weeks thereafter from first dose until disease progression or completion of the study (approximately 2 years)
  Use Investigator tumor measurements to identify objective response rate, duration of response, disease control rate, time to response, and progression free survival.
Pharmacokinetic (PK) measure: area under the concentration-time curve over the dosing interval (AUCtau) | Measured from pre-infusion Cycle 1 to Day 30 post last dose.
  Measure the AXN-2510 concentration in blood as a function of time
Pharmacokinetic (PK) measure: minimum observed serum concentration (Cmin) | Measured from pre-infusion Cycle 1 to Day 30 post last dose.
  Measure the minimum serum concentration of AXN-2510
Pharmacokinetic (PK) measure: maximum observed serum concentration (Cmax) | Measured from pre-infusion Cycle 1 to Day 30 post last dose.
  Measure the maximum serum concentration of AXN-2510
Pharmacokinetic (PK) measure: time at which maximum serum concentration occurs (Tmax) | Measured from pre-infusion Cycle 1 to Day 30 post last dose.
  Measure of time to reach maximum plasma concentration after administration of AXN-2510
Changes in Pharmacodynamic (PD) biomarker sVEGF-A | Measured from pre-infusion Cycle 1 to Day 30 post last dose.
  Activity of free soluble vascular endothelial growth factor A (sVEGF-A) will be assessed
Changes in Pharmacodynamic (PD) biomarker T-cells | Measured from pre-infusion Cycle 1 to Day 30 post last dose.
  Changes in T-cell subtypes will be assessed
To evaluate the immunogenicity of AXN-2510. | Measured from pre-infusion Cycle 1 to Day 30 post last dose.
  Measure the amount of participant antibodies created against AXN-2510.

CONTACTS AND LOCATIONS:
Overall Officials: Jill I Loftiss, RN, Study Director — Instil Bio
Locations (7):
- United States (7):
  - Carolina BioOncology, Huntersville, North Carolina
  - Sarah Cannon Research Institute at Mary Crowley, Dallas, Texas
  - New Experimental Therapeutics (NEXT) Oncology - Houston, Houston, Texas
  - NEXT Houston, Houston, Texas
  - New Experimental Therapeutics of San Antonio - NEXT Oncology, San Antonio, Texas
  - NEXT San Antonio, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
Testing of samples may occur late in the study, and may not be available during patient treatment.